CLINICAL TRIAL: NCT03923517
Title: RHAPSODY-plus: Online Counseling for Family Caregivers of Patients With Young Onset Dementia
Acronym: RHAPSODY-plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Janine Diehl-Schmid, Professor, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RP123
Record Dates: First submitted 2019-04-12; First posted 2019-04-22 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Early Onset Alzheimer Disease; Frontotemporal Dementia
Keywords: Young onset dementia; caregiver; online intervention; online communication technology
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: This pilot study is a single-site study. One intervention group (no control group) Not randomised Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YOD caregiver (Experimental): The participants will be encouraged to use RHAPSODY for four weeks. After that they will have two individual MEET sessions with experts (social worker and psychologist).
  Interventions: Device: RHAPSODY online program and MEET online sessions

INTERVENTIONS:
Device: RHAPSODY online program and MEET online sessions — internet-based information and skill-building program (RHAPSODY) specifically developed for family carers of care recipients with young onset dementia (Kurz, et al., 2016).
  MEET is a software for online meetings.

SUMMARY:
The RHAPSODY-plus project consists of two parts. In a first step carers of people with young onset dementia (YOD; onset before the age of 65) have the opportunity to use the RHAPSODY online program (Kurz et al., 2016) to inform themselves about different topics on young onset dementia. In a second step the participants will receive two individual counseling sessions via MEET (online videoconferencing) with a social worker and a psychologist. Goal is to investigate whether these counseling sessions have an additional benefit.

DETAILED DESCRIPTION:
RHAPSODY-plus is a joint project of the Technische Universität München, Zentrum für kognitive Störungen and the Melbourne University. The project consists of two parts. In a first step carers of people with young onset dementia (YOD; onset before the age of 65) have the opportunity to use the RHAPSODY online program (Kurz et al., 2016) for four weeks. This e-learning program focuses on managing problem behaviors, dealing with role change, obtaining support, and looking after oneself. In a second step the participants will receive two individual counseling sessions via MEET (online videoconferencing). In a first session carers can talk with a social worker about individual problems concerning social, financial and legal issues. In a second session with a psychologist personal and emotional problems can be addressed. These two sessions are about 60 minutes. The study investigates whether these counseling sessions have an additional benefit. The primary aim is to determine whether the intervention is considered acceptable and useful by the participants. Secondary aim is to investigate whether the intervention is feasible. The sample size will be determined when data saturation is reached (no new themes emerge from the qualitative data at the final feedback session). From previous experiences with pilot studies using qualitative methods we expect this to be achieved with approximately 20 participants. This number of participants should also ensure that a diverse group of carers is participating in this pilot study (both genders; different age groups, types of relatives; diagnoses (both FTD and AD) for care recipients; environments (city versus rural); socioeconomic status; and carer stressors (carers with children, carers who hold a job, carers with different stressors, etc.).

ELIGIBILITY:
Inclusion Criteria:

* informal carer of a person with YOD who has been diagnosed with either Frontal Temporal Dementia (FTD) or Alzheimer's Disease (AD) 12 months ago or less;
* the carer has face-to-face contact with the person with YOD at least twice a weak;
* the carer has a working computer and internet access in his home;
* the carer is available for the intervention duration of approximately eight weeks;
* the carer is fluent in German;
* signed consent form.

Exclusion Criteria:

* the carer has face-to-face contact with the person with YOD less than twice a week;
* the person with YOD the carer is caring for has a different dementia cause other than FTD or AD or the diagnosis is older than 12 months;
* the carer does not have a working computer and internet access at home or is not confident to use them;
* the carer is not available for the approximately eight week intervention duration;
* the carer is not fluent in German;
* the carer has a significant health problem or disability, which precludes him/her from participating in the study;
* no signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Acceptability and usefulness | 1 year
  The primary aim of this study is to determine whether the online-video conference-counseling is considered acceptable and useful by the family caregivers. This will be derived from the analysis of caregiver interviews (qualitative research methods).

SECONDARY OUTCOMES:
Feasibility | 1 year
  Secondary aim is to investigate whether the intervention is feasible for the caregivers.This will be derived from the analysis of caregiver interviews (qualitative research methods)

CONTACTS AND LOCATIONS:
Overall Officials: Janine Diehl-Schmid, Prof., Principal Investigator — Technical University of Munich
Locations (1):
- Zentrum für kognitive Störungen, Psychiatrische Klinik und Poliklinik, Klinikum Rechts der Isar, TU München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kurz A, Bakker C, Bohm M, Diehl-Schmid J, Dubois B, Ferreira C, Gage H, Graff C, Hergueta T, Jansen S, Jones B, Komar A, de Mendonca A, Metcalfe A, Milecka K, Millenaar J, Orrung Wallin A, Oyebode J, Schneider-Schelte H, Saxl S, de Vugt M. RHAPSODY - Internet-based support for caregivers of people with young onset dementia: program design and methods of a pilot study. Int Psychogeriatr. 2016 Dec;28(12):2091-2099. doi: 10.1017/S1041610216001186. Epub 2016 Aug 30. PMID 27572272
- [Background] Lautenschlager NT, Diehl-Schmid J, Loi SM, Mayer J, Tensil M, Kurz AF. Modern technology to support carers of care recipients with dementia or functional mental illness: promising progress, but a long road ahead. Int Psychogeriatr. 2017 Dec;29(12):1933-1935. doi: 10.1017/S1041610217002150. PMID 29130870